CLINICAL TRIAL: NCT04401904
Title: Effect of SGLT2 Inhibition on Aging-related Biomarkers in Older Obese Adults With Pre-diabetes
Brief Title: SGLT2 Inhibition in Older Obese Adults With Pre-diabetes
Acronym: SGLT2i
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20190766H; 2P30AG044271 (NIH)
Record Dates: First submitted 2020-04-22; First posted 2020-05-26 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Aging
Keywords: pre-diabetes; aging; glucose metabolism; borderline diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — dapagliflozin; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: 20 completed subjects are planned. Each subject will be randomized to either the experimental group of dapagliflozin 10mg daily for 12 weeks or the control group of nutritional counseling for weight loss.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): 10 participants with pre-diabetes will be randomized to the experimental group to receive dapagliflozin 10mg by mouth daily for 12 weeks.
  Interventions: Drug: Dapagliflozin 10 mg
- Nutritional Counseling (Other): 10 participants with pre-diabetes will be randomized to receive nutritional counseling weekly for 12 weeks
  Interventions: Behavioral: Nutritional counseling

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — 10 participants randomized to receive 12 weeks of daily dapagliflozin 10mg by mouth
  Other Names: Farxiga
  Arms: Dapagliflozin
Behavioral: Nutritional counseling — 10 participants randomized to receive 12 weeks of weekly counseling on nutrition
  Arms: Nutritional Counseling

SUMMARY:
Inhibitors of the sodium-glucose co-transporter (SGLT2) are FDA-approved for the treatment of type 2 diabetes (T2DM). Their mechanism of action involves lowering of blood glucose concentration secondary to increased glucose excretion of glucose by the kidney. These drugs also improve body weight, blood pressure, and cardiac function. Based on these pleiotropic effects, including its calorie restriction-mimetic properties, the study team hypothesize that SGLT2 drugs will impact several basic aging-related processes, including reductions in oxidative damage to DNA and proteins, advanced glycation end products (AGE) and receptor for AGE (RAGE), cellular senescence, and mitochondrial function.

DETAILED DESCRIPTION:
Investigations into the aging process have identified major cellular dysfunctions that contribute to aging, including but not limited to increased burden of damaged DNA and protein, reduction in mitochondrial respiration, and the development of pro-inflammatory senescent cells. Developing and testing interventions that interact with multiple points of this spectrum may delay the aging process. Based on prior investigations, the study team believe the SGLT2 inhibitor class of drugs may target these basic mechanisms involved in the aging process and propose testing in a high-risk human population to evaluate their effectiveness in ameliorating aging-associated dysfunctions. Specifically, the investigators hypothesize that SGLT2i drugs will lead to reductions in oxidative damage to DNA and proteins, AGE-RAGE, and cellular senescence, which will be accompanied by improvements in mitochondrial function. If the hypothesis is correct, these findings could lead to the development of new approaches to increase both health-span and lifespan.

This is a single center, open-label, randomized controlled trial. The target enrollment for this pilot study is 20 completed subjects, split evenly between experimental and control groups. Each subject will be randomized to either the experimental group of dapagliflozin 10mg daily for 12 weeks or the control group of nutritional counseling for weight loss. Health-span and clinical evaluations will be taken at baseline and at weeks 10-12 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or post-menopausal women.
2. Age= 60+ years.
3. All ethnic groups.
4. Body Mass index (BMI) between 30-38 kg/m2.
5. Diagnosis of pre-diabetes (HbA1c 5.7-6.4% and 2 hr. Oral Glucose Tolerance Test (OGTT) glucose between 140-199 mg/dL, evaluated at Visit 1 and 2).
6. Stable body weight (±3% for ≥3 months).
7. Willing to adhere to medication regimen for three months.
8. Montreal Cognitive Assessment score ≥21

Exclusion Criteria:

1. Diagnosis of diabetes based on American Diabetes Association (ADA) criteria
2. Impaired renal function with estimated Glomerular Filtration Rate (eGFR) < 45 mL/min/1.73m2 .
3. Impaired liver function with labs ≥3 times upper limits of normal range
4. Abnormal hematocrit with lower limits of ≤30%
5. Abnormal triglycerides with upper limits ≥600 mg/dL
6. Abnormal Thyroid stimulating hormone (TSH) values ≤0.3 and ≥10
7. Urinalysis results with ˃ 5-10 white blood cell count
8. Concomitant medications known to affect glucose and lipid homeostasis (anti-diabetes medications, glucocorticoids, atypical antipsychotics, anti-transplant rejection medications, anti-retrovirals).
9. Current treatment with anticoagulants (warfarin). Aspirin (up to 325 mg) and clopidogrel will be permitted if these can be held for seven days prior to the biopsies.
10. History of recent cardiovascular event in the last 6 months or Heart Failure (New York Heart Classification greater than class III-IV; recent EKG changes that suggest active heart disease
11. Poorly controlled blood pressure (systolic BP>180, diastolic BP>100 mmHg).
12. Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, and uncontrolled psychiatric disease (Subjects with depression, anxiety, PTSD, etc. can enroll if controlled and on stable medication)
13. Blood donation within 2 months prior to enrollment
14. History of frequent UTI

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Solis-Herrera, Principal Investigator — University of Texas Health at San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Protocol, Statistical Analysis Plan, Published data
Supporting Information: Study Protocol, SAP
Time Frame: After study completion, upon publication of data and on ClinicalTrials.gov 1 year after primary completion date of study.
Access Criteria: Data will be analysed by a statistician for publication and by direct communication with the principal investigator

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Nutritional Counseling
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Nutritional Counseling | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 8 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: AGE-RAGE Measurement in Plasma
Description: Change in AGE-RAGE measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Dapagliflozin | Nutritional Counseling
Number analyzed (Participants) | 10 | 10
pg/mL | -172 (121) | -86 (112)

2. Secondary Outcome: Grip Strength
Description: Change in grip strength measured using a hand-held dynamometer in Newton meters (Nm)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Error); unit: Nm
Arm/Group | Dapagliflozin | Nutritional Counseling
Number analyzed (Participants) | 10 | 10
Nm | -2 (1.3) | -1 (1.2)

3. Secondary Outcome: 6 Minute Walking Distance
Description: Change in walking distance in the 6 minute walking test.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Error); unit: m
Arm/Group | Dapagliflozin | Nutritional Counseling
Number analyzed (Participants) | 10 | 10
m | 6.6 (7.6) | 9.1 (11.8)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Dapagliflozin | Nutritional Counseling
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT04401904/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT04401904/ICF_001.pdf